CLINICAL TRIAL: NCT06305546
Title: Comparison Of Different Antiplaque Agents On Gingivitis In Patients Undergoing Fixed Orthodontic Treatment: A Double-Blind, Randomized Controlled Trial.
Brief Title: Comparisons Of Different Antiplaque Agents On Gingivitis In Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anam Sattar (Other)
Responsible Party: Sponsor-Investigator, Anam Sattar, Senior Registrar, Department of Orthodontics, Principal Investigator., Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2911
Record Dates: First submitted 2023-12-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gingivitis
Keywords: gingivitis,; fixed orthodontic treatment,; anti plaque gels
MeSH Terms: conditions — Gingivitis | interventions — chlorhexidine gluconate; Metronidazole; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The trial was a double blinded (patients and investigators). We were helped from a member of our department who is not a part of the study, to transfer the gels from commercial tubes to blank containers. The randomization codes remained unknown until data analysis was completed. Randomization was done by computer-generated software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- group A (Experimental)
  Interventions: Drug: Chlorhexidine Gluconate
- GROUP B (Experimental)
  Interventions: Drug: Metronidazole
- GROUP C (Experimental)
  Interventions: Drug: combination gel (chlorhexidine and metronidazole)
- GROUP D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — For two weeks, all individuals were instructed to use pea-sized gel on their gingiva two times a day. To ensure patient compliance, we assigned patients with log sheets to fill daily on whether they used the gel consistently every day twice a day for 2 weeks. Patients were also instructed to return the container of gel on the day of follow-up.
  Other Names: CHX
  Arms: group A
Drug: Metronidazole — For two weeks, all individuals were instructed to use pea-sized gel on their gingiva two times a day. To ensure patient compliance, we assigned patients with log sheets to fill daily on whether they used the gel consistently every day twice a day for 2 weeks. Patients were also instructed to return the container of gel on the day of follow-up.
  Arms: GROUP B
Drug: combination gel (chlorhexidine and metronidazole) — For two weeks, all individuals were instructed to use pea-sized gel on their gingiva two times a day. To ensure patient compliance, we assigned patients with log sheets to fill daily on whether they used the gel consistently every day twice a day for 2 weeks. Patients were also instructed to return the container of gel on the day of follow-up.
  Arms: GROUP C
Drug: Placebo — For two weeks, all individuals were instructed to use pea-sized gel on their gingiva two times a day. To ensure patient compliance, we assigned patients with log sheets to fill daily on whether they used the gel consistently every day twice a day for 2 weeks. Patients were also instructed to return the container of gel on the day of follow-up.
  Arms: GROUP D

SUMMARY:
Fixed orthodontic treatment affects the periodontium by allowing plaque accumulation on teeth if the oral ecosystem is unfavorable which initially causes gingivitis to progress into periodontitis, and later enamel demineralization occurs. Yáñez-Vico et al observed that regular modifications per checkups were painful and unpleasant for the patient thus the patients undergoing fixed orthodontic treatments compromised their oral hygiene. This creates plaque retention sites which can lead to developing white spot lesions, caries, and periodontitis

DETAILED DESCRIPTION:
Metal brackets were used on the teeth such as incisors, canines, and premolars as well as bands on the 1st molars to treat all patients with the same kind of orthodontic appliances. Metal Brackets were bonded by the principal investigator with the direct bonding technique by using light cure adhesives. General oral hygiene instructions were given by the clinician to each participant in the study.

Participants were divided into four groups through computer-generated software. Group A participants used 1% metronidazole gel, Group B participants used 0.25% chlorhexidine gel. Group C participants used a combination gel (1% Metronidazole and 0.25% Chlorhexidine). Group D participants used a placebo gel. All participants were instructed to follow oral hygiene measures such as brushing twice a day with a soft brush with fluoridated toothpaste, and use of floss or interdental brushes. For two weeks, all individuals from groups A, B, C, and D were instructed to use pea-sized gel on their gingiva two times a day. To ensure patient compliance, the investigators assigned patients with log sheets to fill daily on whether they used the gel consistently every day twice a day for 2 weeks. Patients were also instructed to return the container of gel on the day of follow-up.

OUTCOMES:

The primary outcome included the measurement of indices during study time from baseline (T0) to 2weeks (T1), 4 weeks (T2), 8 weeks (T3) and 12 weeks(T4) . The investigators have evaluated Gingival Index and Bleeding Index by probing and assessing the gingiva and Orthodontic Plaque index by plaque disclosing tablets, and examined six standard sites on incisors, canine, and premolars as described by Gettinger et al. Banded first molars were not included because banding itself can compromise periodontal health. The study sites were assessed by using CPITN probe. Six proximal line angles were investigated for gingivitis on the selected teeth: Right maxillary second premolar, mesiobuccal line angle; right maxillary canine, distobuccal line angle; left maxillary central incisor, distopalatal line angle; right mandibular central incisor, distolingual line angle; left mandibular canine, distobuccal line angle; left mandibular second premolar, mesiobuccal line angle.

If any of the study teeth were missing, then the corresponding tooth on the opposite side was evaluated.

Patients were only included in the trial if they have Gingival index, Orthodontic plaque index scores ≥2 and Bleeding index ≥ 1 on any three or more than three of the six teeth that were examined in the study. The total combined GI and BI indexes were computed by averaging the measured values at T0, T1, T2, T3 and T4 . For OPI, the score was calculated by counting the number of teeth with plaque accumulation at each time interval.

ELIGIBILITY:
Inclusion Criteria

* Patients between the ages of 16 - 35 years with moderate to severe crowding and receiving fixed orthodontic treatment for at least six months were eligible.
* Patients with gingival, and ortho plaque indices ≥ 2 and bleeding index ≥ 1 were also included in the inclusion criteria.

Exclusion criteria include

* systematically unhealthy patients with comorbidities such as blood dyscrasias, rheumatic fever, congenital heart disease, and diabetes mellitus.
* Smokers
* participants who show no motivation to take care of their teeth,
* people with disabilities who are physically dependent in any way.
* Patients with allergies to chlorhexidine and metronidazole,
* women who are pregnant or lactating.
* Patients with clinical attachment loss and calculus.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
gingival index | 12 weeks
  Gingival index Score 0: no inflammation Score 1: Mild inflammation of gingiva. No bleeding on probing. Score2: Moderate inflammation, Red, edematous and shiny gingiva, bleeding on probing.
  Score 3: Severe inflammation, Red, edematous and ulcerated gingiva. There is spontaneous bleeding
bleeding index | 12 weeks
  Bleeding Index Score 0: absence of bleeding after 30 seconds Score 1: presence of bleeding after 30 seconds Score 2: immediate bleeding
orthodontic plaque index | 12 weeks
  Orthodontic Plaque Index 0: No plaque deposits on the tooth surfaces surrounding the bracket base
  1. Plaque deposits on one tooth surface at the bracket base
  2. Plaque deposits on two tooth surfaces at the bracket base
  3. Plaque deposits on three tooth surfaces at the bracket base
  4. Plaque deposits on four tooth surfaces at the bracket base

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided